CLINICAL TRIAL: NCT02967770
Title: A Randomized Phase II Trial Comparing Molecularly Tailored Therapy to Physician's Discretion Standard of Care as Second-Line Therapy for Patients With Metastatic Pancreatic Cancer
Brief Title: Molecularly Tailored Therapy to Standard of Care as Second-Line Therapy in Metastatic Pancreatic Cancer
Acronym: PanCAN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Issues with patient recruitment.
Sponsor: Georgetown University (Other)
Collaborators: Thomas Jefferson University (Other); Sinai Health System (Other); Virginia Mason Hospital/Medical Center (Other); Cedars-Sinai Medical Center (Other); George Mason University (Other); Caris Life Sciences (Industry); Theranostics Health, Inc (Unknown); Guardant Health, Inc. (Industry); Companion Diagnostics, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1120
Record Dates: First submitted 2016-11-02; First posted 2016-11-18 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Metastatic; Pancreas; Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Molecularly Tailored Therapy (Experimental): Patients will be treated according to their molecular profile and accordingly, the 29 evaluable patients enrolled may receive one of a dozen, or dozens of treatment regimens.
  Interventions: Other: Molecularly Tailored Second Line Therapy
- Physician's Discretion Standard of Care (Active Comparator): Patients will be treated according to physician discretion standard of care regimen.
  Interventions: Drug: Standard of Care Second Line Therapy

INTERVENTIONS:
Other: Molecularly Tailored Second Line Therapy — This trial is designed to assess the efficacy of MTT vs. SOC therapy as second-line therapy in patients with metastatic pancreatic cancer.
  Arms: Molecularly Tailored Therapy
Drug: Standard of Care Second Line Therapy
  Arms: Physician's Discretion Standard of Care

SUMMARY:
The purpose of this study is to determine whether molecularly tailored therapy can improve the efficacy of treatment when compared to standard chemotherapy combinations for patients with metastatic pancreatic cancer receiving their second line of therapy for metastatic disease.

DETAILED DESCRIPTION:
This is an open label, randomized Phase II trial for patients with metastatic pancreatic cancer. The trial is designed to compare the outcomes (primary endpoint will be progression-free survival (PFS)) for patients who receive molecularly-tailored therapy (MTT) to those who receive physician discretion standard of care (SOC). To successfully allow for this assessment, and minimize confounding variables, we will need to ensure that:

* There is enough tissue for the molecular profiling to occur. Thus, only patients with adequate tumor tissue will be allowed to enroll.
* There is enough time for the molecular profiling to be completed; for the medical review panel (MRP) to render a determination on the optimal molecularly-guided therapy; and for the treating physician to obtain access to therapies, particularly if the MRP-determined therapy includes an off-label treatment OR a clinical trial. We anticipate this process will take a minimum of 4 weeks.

These factors will inevitably lead to a selection bias towards patients with a better prognosis. However, the randomization design should mitigate this selection bias.

Patients with metastatic pancreatic cancer who are actively on (or about to initiate) first-line therapy, who meet the inclusion and exclusion criteria as detailed in Section 3 will be enrolled. For all enrolled patients, at the time of enrollment, the treating physician will be asked to submit the planned second line SOC treatment he/she would recommend.

In an effort to streamline accrual, and based on data that demonstrate that the tumor genetic profile does not change significantly overtime in patients with pancreatic cancer, archived tumor tissue may be used for determination of MTT. The archived tissue may be, for example, core needle biopsies obtained at the time of establishing the diagnosis of metastatic disease; or for example, a surgical specimen obtained prior to the identification of metastatic disease. Archived tissue may be used as long as there is sufficient tissue for full molecular testing. Of note, even if sufficient archived tissue is available for testing, patients will still be required to undergo a new biopsy to obtain fresh tissue for ex vivo analysis, prior to initiation of second line therapy.

Patients will then undergo tumor testing, as detailed next. If a patient undergoes tumor testing but his/her disease progresses on first-line therapy prior to an MRP-determined therapeutic plan, then the patient will be considered a screen failure, and will be replaced.

Then, for all patients for whom adequate tissue is available for profiling, an MRP-determined therapeutic plan will be developed. This process of determining the MRP-determined therapeutic plan will be kept blinded to the treating physician (i.e. each treating physician will NOT be involved in the determination of MTT for his/her patient) - but once the plan is available, the patients will be randomized to either MTT or SOC (See Figure 4):

Patients will be monitored closely while on first-line therapy. For patients who are randomized to MTT, the MRP-determined therapeutic plan will be unblinded to the treating physician, and preparation for MTT can begin, including acquiring access to off label therapy, if required. Patients who are randomized to SOC therapy will receive the SOC treatment initially recommended by the treating physician

Once a patient experiences disease progression on first-line therapy, they will receive MTT vs. SOC as second-line therapy, according to their randomization. Patients in both groups will receive second-line therapy until disease progression or therapy intolerance (with dose and schedule modifications as needed). Response assessment will occur approximately every 8 weeks (based on the calendar) as determined from the time of the initiation of therapy. All patients will have the option to undergo a repeat tumor biopsy upon disease progression.

Once patients on SOC therapy experience progressive disease on second-line therapy, the MRP-determined therapeutic plan will unblinded to the treating physician, and MTT therapy can be administered as third-line therapy (crossover to MTT). Third-line therapy can also incorporate correlative analyses on the patient tumor samples tested ex vivo (detailed below) if these results are available at the time that third line therapy is required. As this may impact the overall survival assessment, the primary endpoint is disease progression at 4 months (PFS4mos), and the primary objective is to compare the PFS4mos for MTT treated vs. SOC treated patients. We hypothesize that MTT will improve the PFS4mos from 50% for SOC (based on historical data), to ≥75%. We anticipate having 80% power to detect an improvement in the PFS4mos from 50% to ≥75% (hazard ratio (HR) = 0.5), assuming a 1-sided significance level of 0.05 and an accrual rate of 4 patients per month (see statistics below).

Of note, the treating physician may opt to incorporate the molecular data to select third-line therapy for patients whose disease progresses on second-line MTT therapy. The results of ongoing analyses and testing of the patient tumor samples, ex vivo including the CRCs, organoids, and the zebrafish avatars may be available at the time that the patient requires third-line therapy. If so, the treating physician may incorporate the results of these analyses into the decision plan for third-line therapy. These patients will continue to be followed longitudinally for survival, but there will be no formal comparison of third line therapy outcomes with the "crossover" group.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic adenocarcinoma of the pancreas (at enrollment)
2. Actively on (or about to initiate) first line therapy for metastatic pancreatic cancer (at enrollment)

   * Patients may have had neo-adjuvant and/or chemotherapy that must have been completed >3 months prior to starting first line therapy
   * Patients may be actively on "maintenance" therapy, such as maintenance capecitabine up to starting first line therapy for metastatic disease
3. Radiographically measurable disease (prior to initiation of second-line therapy)
4. Tumor deposits that are clearly accessible for serial tumor biopsies - A patient's biopsied lesion must be at least 1cm in diameter (in at least one dimension) (prior to initiation of second-line therapy)
5. Age ≥ 18 years (at enrollment)
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Table 6, Appendix D) (at enrollment)
7. Adequate hepatic, bone marrow, and renal function at the time of enrollment AND at initiation of second line therapy:

   * Bone Marrow: Absolute neutrophil count (ANC) ≥ 1,500/mm3; Platelets ≥ 75,000/mm3; Hemoglobin ≥ 9.0 g/dL
   * Patients may have a transfusion of red blood cells to meet the hemoglobin requirement
   * Renal function: Serum creatinine ≤ 1.5 X upper normal limit of institution's normal range OR creatinine clearance ≥ 50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal
   * Hepatic function: Aspartate transaminase (AST) and Alanine transaminase (ALT) ≤ 3 X the upper normal limit of institution's normal range; bilirubin ≤ 1.5 X the upper limit of normal. For patients with known hepatic metastases, AST and ALT ≤ 5 X the upper normal limit of institution's normal range
   * Prothrombin Time and Partial Thromboplastin Time (PTT) must be ≤ 2 X the upper limit of the institution's normal range and International Normalized Ratio (INR) < 2. Subjects on anticoagulation (such as coumadin) will be permitted to enroll as long as the INR is in the acceptable therapeutic range as determined by the investigator
8. Patients must have fully recovered from all effects of surgery (prior to initiation of second-line therapy). Patients must have had at least two weeks after minor surgery and four weeks after major surgery before starting therapy. Minor procedures requiring "Twilight" sedation such as endoscopies or mediport placement may only require a 24-hour waiting period, but this must be discussed with an investigator.
9. Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to initiation of treatment and/or postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential (at enrollment).
10. Subject is capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consent, approved by the Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures (at enrollment).

Exclusion Criteria:

1. Known or suspected brain or central nervous system metastases, irrespective of prior treatment
2. The subject has had another active malignancy within the past three years except for cervical cancer in situ, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin. Questions regarding the inclusion of individual subjects should be directed to the Study Chair.
3. Clinically significant peripheral neuropathy at the time of enrollment (defined in the NCI Common Terminology Criteria for Adverse Events Version 4.0 [CTCAE v4.0] as grade 2 or greater neurosensory or neuromotor toxicity)
4. Patients receiving any other investigational agents.
5. Active severe infection, or known chronic infection with HIV or hepatitis B virus

   -Patients with chronic Hepatitis C virus may be enrolled if there is no clinical/laboratory evidence of cirrhosis AND the patient's liver function tests fall within the parameters set in Section 3.2.7.3, Inclusion Criteria, Hepatic function
6. Cardiovascular disease problems including unstable angina, therapy for life-threatening ventricular arrhythmia, or myocardial infarction, stroke within the last 3 months, or a diagnosis of congestive heart failure
7. Life-threatening visceral disease or other severe concurrent disease
8. Women who are pregnant or breastfeeding
9. Anticipated patient survival under 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
4 month progression free survival rate | 4 months after treatment start
  4 month progression free survival rate (PFS4mos) of MTT vs. SOC therapy as second line therapy in patients with metastatic pancreatic cancer

SECONDARY OUTCOMES:
Median overall survival | 60 months
Objective Response Rate | 60 months
Disease control rate | 6 months
  Disease Control Rate (DCR) = Complete Response (CR)+ Partial Response (PR) + Stable Disease (SD) at 6 months
Median progression-free survival | 60 months
Change in tumor marker levels | 60 months
  Cancer Antigen (CA) 19-9 or Carcinoembryonic antigen (CEA)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pishvaian, MD, PhD, Study Chair — Georgetown Lombardi Comprehensive Cancer Center
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tesfaye AA, Wang H, Hartley ML, He AR, Weiner L, Gabelia N, Kapanadze L, Shezad M, Brody JR, Marshall JL, Pishvaian MJ. A Pilot Trial of Molecularly Tailored Therapy for Patients with Metastatic Pancreatic Ductal Adenocarcinoma. J Pancreat Cancer. 2019 May 2;5(1):12-21. doi: 10.1089/pancan.2019.0003. eCollection 2019. PMID 31065624